CLINICAL TRIAL: NCT02802644
Title: A Prospective, Multi-center, Randomized, Controlled Study to Evaluate the Effect of DiPeptidyl-Peptidase 4 Inhibitor on Vascular Healing After Biodegradable Polymer Based Sirolimus Eluting Stent Implantation in Diabetic Patients: OCT Study (DIAMOND-OCT)
Brief Title: The Effect of DPP4 Inhibitor on Vasclular Healing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University (Other)
Responsible Party: Principal Investigator, Sang-Wook Kim, MD, PhD, Chung-Ang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAU001
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Acute Coronary Syndrome; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Acute Coronary Syndrome; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DPP-4 Inhibitor (Experimental): Any dose of Sitagliptin for 6 months with any other oral anti-diabetic medication
  Interventions: Drug: Sitagliptin
- Non DPP-4 Inhibitor (Active Comparator): Oral anti-diabetic medication except DPP-4 inhibitor
  Interventions: Drug: Non DPP-4 Inhibitor

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin is indicated to control hyperglycemia in type 2 diabetic patients.
  Other Names: Janiuvia
  Arms: DPP-4 Inhibitor
Drug: Non DPP-4 Inhibitor — This group patients is permitted to take any other oral anti-hyperglycemic agents except sitagliptin.
  Arms: Non DPP-4 Inhibitor

SUMMARY:
This study evaluate the effect of dipeptidyl-peptidase 4 inhibitor on vascular healing after biodegradable polymer based sirolimus eluting stent implantation in diabetic pateints.

ELIGIBILITY:
Inclusion Criteria:

* Non-ST segement elevation acute coronary syndrome

Exclusion Criteria:

* Left main disease
* Known hypersensitivity or contraindication to any of the following medications: Heparin, aspirin, clopidogrel, sirolimus, siptagliptin and statin
* Congestive heart failure (patients with LVEF <30% or cardiogenic shock)
* Uncontrolled myocardial ischemia (repeated chest pain or dyspnea after revascularization)
* Uncontrolled ventricular arrhythmia
* History of malignancy with chemotherapy
* Serious hematologic disease (e.g. CML, MDS)
* Current infectious disease needs antibiotics therapy
* Creatinine level >1.5 mg/dL or dependence on dialysis
* Other severe concurrent illness (e.g. active infection, malignancy).
* Life expectancy of less than one year
* Pregnancy or women with potential childbearing
* Type I DM
* Treatment with insulin
* History of pancreatitis
* Who cannot read the informed consent form (e.g. illiteracy, foreigner)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Neointimal coverage assessed by optical coherence tomography | 6 months

SECONDARY OUTCOMES:
Malapposition, neointimal thickness or any optical coherence tomographic finding | 6 months
Biomarkers | 6 months
  CD 34+ cell, hs CRP ect.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Wook Kim, MD, PhD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (6):
- South Korea (6):
  - Keimyung University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Jeju National University Hospital, Jeju City
  - Chung-Ang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon